CLINICAL TRIAL: NCT06736600
Title: Patient-identified Values as Outcome Targets (PIVOT) Feasibility Pilot Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024-1305; NCI-2024-10309 (Other: Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2024-12-12; First posted 2024-12-17 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Peripheral Neuropathy Due to Chemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Goal Encouragement (Experimental): Eligible participants will be identified using electronic health record
  Interventions: Behavioral: Goal Attainment Scaling (GAS)
- No Goal Encouragement (Experimental): Eligible participants will be identified using electronic health record
  Interventions: Behavioral: Goal Attainment Scaling (GAS)

INTERVENTIONS:
Behavioral: Goal Attainment Scaling (GAS) — Goal-setting tele-coaching and the well-studied Patient Priorities Care framework will assist participants with bothersome CIPN identify their most important health goals and scale them into specific, measurable, achievable, relevant, and time-bound (SMART) goals

SUMMARY:
A behavioral trial aimed at helping patients identify what matters most to them and is part of a larger effort to pivot from disease-oriented care to whole-person care.

DETAILED DESCRIPTION:
Primary Objectives:

The primary objective of the pilot clinical trial is to evaluate feasibility, operationalized as attrition, acceptability, and adherence rates of the GAS measure.

Secondary Objectives:

To evaluate initial efficacy across both arms (pre-post comparison) and between arms (A-B comparison) of goal encouragement. Due to the pilot nature of this work and a lack of published effect size estimates, this trial is unlikely to be adequately powered to estimate true efficacy. However, this trial will provide a rich source of preliminary data and effect size estimates that can be utilized to conduct formal power analysis for a larger efficacy trial.

The tertiary objective will be to identify themes within the GAS measures created by participants, utilizing grounded theory inductive coding of themes into broader categories, and comparing against the common categories pre-identified within the Patient Priorities Care framework.

The quaternary objective will be to assess a novel measure of CIPN outcomes called the Individual Neuropathy Report Card against current common CIPN measures.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated electronic informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Age 18 or older.
* Documented diagnosis of chemotherapy-induced peripheral neuropathy meeting the following criteria: 1) onset associated with timing of neurotoxic chemotherapy and 2) symptomatic reports of peripheral neuropathy.
* Access to smartphone and internet for participating in a technology-based intervention
* Upcoming in-person appointment in the Main Hospital Pain Management Clinic 4-6 weeks from the consent date.
* English-speaking
* Pain or bothersome symptoms present most days of the week at an average of ≥4/10 on the Numeric Rating Scale for the past 3 months
* No longer receiving cancer treatment or has been on stable maintenance treatment for the past 3 months.
* Resides in the Houston Metroplex
* A score ≤7 on the validated Six Item Cognitive Impairment Test (6CIT) for unimpaired cognition

Exclusion Criteria:

* Provision of signed and dated electronic informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Age 18 or older.
* Documented diagnosis of chemotherapy-induced peripheral neuropathy meeting the following criteria: 1) onset associated with timing of neurotoxic chemotherapy and 2) symptomatic reports of peripheral neuropathy.
* Access to smartphone and internet for participating in a technology-based intervention
* Upcoming in-person appointment in the Main Hospital Pain Management Clinic 4-6 weeks from the consent date.
* English-speaking
* Pain or bothersome symptoms present most days of the week at an average of ≥4/10 on the Numeric Rating Scale for the past 3 months
* No longer receiving cancer treatment or has been on stable maintenance treatment for the past 3 months.
* Resides in the Houston Metroplex
* A score ≤7 on the validated Six Item Cognitive Impairment Test (6CIT) for unimpaired cognition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-04-18 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse Events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Alice Ye, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M. D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org